CLINICAL TRIAL: NCT05904652
Title: A Randomised, Feasibility Trial of Simultaneous Application of Flow at Extubation (SAFEx) in Patients Requiring Intubation and Ventilation for the Management of Acute Respiratory Failure
Brief Title: High Flow Nasal Oxygen at Extubation for Adults Requiring a Breathing Tube for Treating Severe Breathing Difficulties
Acronym: Pre-SAFEx
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: Fisher and Paykel Healthcare (Industry); LINET (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GN23CC122
Record Dates: First submitted 2023-05-31; First posted 2023-06-15 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-11

CONDITIONS: Respiratory Insufficiency
Keywords: Extubation Failure; Airway Extubation; Oxygen Inhalation Therapy; Electric Impedance
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Intervention Model Description: Participants will be randomised in a 1:1 manner between two treatments at time of extubation: SAFEx treatment or standard care.
Masking Description: Participants will be randomised in a 1:1 manner using a computer-generated 30 number sequence of '1s' and '2s' from https://www.random.org/ between 1) SAFEx treatment and 2) standard care. A clinician, not involved in the study, will obtain this 30 number sequence and conceal its order within 30 sealed, opaque, numbered envelopes. The investigators will be blinded to the participant's allocation until they have been enrolled in the study, after which the next envelope in the sequence will be opened and treatment allocation will be unblinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SAFEx (Experimental): Electrical Impedance Tomography recording is commenced 15 minutes prior to planned extubation. High Flow Nasal Therapy (HFNT) is commenced at least 10 minutes prior to planned extubation. At 5 minutes before extubation, the flow rate of HFNT should be established at 60 litres per min (or as high as can be tolerated by the participant) and the fraction of inspired oxygen (FiO2) set at 40 percent. Prior to extubation, endotracheal, infraglottic and supraglottic suctioning are performed. Then, the cuff is let down followed by immediate extubation with simultaneous application of HFNT. 10 minutes after extubation, the FiO2 is weaned in a protocolised manner to 21 percent - or as close to 21 percent as possible over 25 minutes. If the participant is safely weaned onto room air, the flow rate of HFNT is then reduced in a protocolised manner over 120 minutes: 60 minutes at 60 litres per minute (or the highest flow rate tolerated) and then 60 minutes at 30 Litres per minute.
  Interventions: Device: Fisher and Paykel "HealthCare Airvo™ 3" high flow system
- Standard Care (Active Comparator): Electrical Impedance Tomography recording commenced 15 minutes prior to planned extubation. Prior to extubation, endotracheal, infraglottic and supraglottic suctioning are performed. Then, the cuff is let down followed by immediate extubation on to low flow conventional oxygen with a fraction of inspired oxygen of up to 40 percent. Then, the participant is weaned at the discretion of their clinician over the next 2 hours and 35 minutes.
  Interventions: Device: Conventional Oxygen Therapy

INTERVENTIONS:
Device: Fisher and Paykel "HealthCare Airvo™ 3" high flow system — High Flow Nasal Oxygen Delivery Device
  Arms: SAFEx
Device: Conventional Oxygen Therapy — Low flow oxygen delivery device (Flow rate between 2 litres per minute and 15 litres per minute)
  Arms: Standard Care

SUMMARY:
The goal of this feasibility study is to learn whether a new approach to breathing tube removal within the Intensive Care Unit is safe and acceptable to participants who require a breathing tube for the management of severe breathing difficulties. The main questions it aims to answer are:

* What is the recruitment rate to the study over 12 months?
* Is the study design acceptable and safe to participants?

Participants will receive high flow nasal oxygen before their breathing tube is removed. The investigators will compare this with standard practice of applying conventional, low-flow oxygen after the breathing tube removed to see if this effects the rate of repeat breathing tube insertion.

The investigators hypothesise that they will recruit 30 participants to the study protocol (15 participants in each group) over 12 months and that our study protocol will be tolerable and acceptable to participants.

ELIGIBILITY:
Inclusion Criteria:

* Participant aged 18 to 80 years old at time of recruitment to study)
* Ventilated for greater than or equal to 48 hours with respiratory failure
* Treating clinician agrees ready for a planned extubation (but pressure support ventilation, fraction of inspired oxygen less than or equal to 40 , positive end expiratory pressure less than or equal to 10 centimetres of water, Respiratory rate less than 20 breaths per minute)
* Minimal secretions
* Neurologically intact (In the opinion of the treating clinician, the participant is unlikely to fail extubation due to their neurological status)
* Cardiovascularly stable (systolic blood pressure greater than or equal to 70 millimetres of mercury, heart rate less than or equal to 150 beats per minute)
* Written informed consent

Exclusion Criteria:

* Cardiac Implant Device
* Internal Neurostimulator
* Unstable Spinal Fracture or Spinal Cord Injury
* Body Mass Index >50kg/m^2
* Skin lesions or dressings over electrode belt site
* Pregnancy or Lactating
* Intercostal Chest Drain (at treating clinician's discretion)
* Severe type II respiratory failure (arterial partial pressure of carbon dioxide greater than or equal to 12 kilopascals)
* Severe acidosis (Hydrogen ion concentration greater than or equal to 80 nanomoles per litre)
* Chronic respiratory disease limiting functional capacity (MRC breathlessness grade IV or V)
* Severe heart failure (New York Heart Association Grade III or IV)
* Decreased GCS
* Cardiovascular instability (systolic blood pressure less than or equal to 69 millimetres of mercury or heart rate greater than or equal to 151 millimetres of mercury )
* Pulmonary embolism
* Nasal obstruction
* Previous bleomycin administration
* Base of skull fracture
* Life expectancy less than or equal to 3 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-09-07 (Actual); Primary Completion 2024-09-07 (Estimated); Study Completion 2024-09-07 (Estimated)

PRIMARY OUTCOMES:
The recruitment rate to the study over 12 months with 1:1 randomisation of participants between SAFEx treatment and standard care. | 12 months
  The associated end point will be the average rate of recruitment per month over 12 months of participants who complete the full study protocol (with a set upper limit of 30 participants recruited to the protocol over 12 months corresponding to a recruitment rate of 2.5 participants per month).

SECONDARY OUTCOMES:
The incidence of Adverse Events and Serious Adverse Events associated with trial procedures. | 72 hours
  This will focus primarily on aspects of SAFEx and Electrical Impedance Tomography Measurement.
Patient Visual Analogue Scale scores for questions exploring the tolerability of SAFEx treatment compared with that of standard care. | 72 hours
  Questions will ask participants to rate their experience on a 1 to 10 scale for:
  * Overall comfort
  * Perceived dyspnoea
  * Ability to speak
  * Ability to hear
  * Ability to clear secretions
  * Sensation of bloating
  * Sensation of dry mouth
  * Sensation of nasal dryness
  * Fear
Withdrawal rate from the study. | 72 hours
  The number of participants requesting to withdraw from the study due to inability to tolerate the trial procedures.
The rate of completion of the SAFEx weaning protocol. | 2 hours 50 minutes
  The percentage of participants who completed the weaning protocol without breaching any of the physiological participant safety criteria.
The duration of weaning tolerated before desaturation occurred. | 2 hours 50 minutes
  The average fraction of inspired oxygen and oxygen flow rate administered in each group before desaturation occurred.
The failure rate of Electrical Impedance Tomography measurement. | 2 hours 50 minutes
  Defined as the proportion of participants in whom impedance data cannot be computed.
The participant self-rated Visual Analogue Scale score for questions exploring the tolerability of Electrical Impedance Tomography Measurement. | 72 hours
  Questions will ask participants to rate their experience on a 1 to 10 scale for:
  * Overall comfort whilst wearing EIT
  * Overall comfort on removal of EIT
  * Overall ease of breathing with EIT
The change in global electrical impedance between each group. | 2 hours 50 minutes
  The change in end expiratory lung impedance and delta impedance between each group.
The reintubation rate in each group. | 72 hours
  The rate of repeat intubation will be measured in each group at 24, 48 and 72 hours post-extubation.

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm AB Sim, MBChB, MD, FRCP, FRCA, FFICM, Principal Investigator — NHS Greater Glasgow and Clyde
Locations (1):
- Department of Critical Care Medicine, Queen Elizabeth University Hospital, Glasgow, Scotland, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymised, processed Physiological, EIT and Questionnaire Data that underlies the results reported in this study will be be made available . Raw data will not be shared.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 5 years following article publication
Access Criteria: Appropriate request made through Enlighten Data Repository (doi will be provided in future publication)

REFERENCES:
- [Background] Rothaar RC, Epstein SK. Extubation failure: magnitude of the problem, impact on outcomes, and prevention. Curr Opin Crit Care. 2003 Feb;9(1):59-66. doi: 10.1097/00075198-200302000-00011. PMID 12548031
- [Background] Krinsley JS, Reddy PK, Iqbal A. What is the optimal rate of failed extubation? Crit Care. 2012 Feb 20;16(1):111. doi: 10.1186/cc11185. PMID 22356725
- [Background] Frutos-Vivar F, Esteban A, Apezteguia C, Gonzalez M, Arabi Y, Restrepo MI, Gordo F, Santos C, Alhashemi JA, Perez F, Penuelas O, Anzueto A. Outcome of reintubated patients after scheduled extubation. J Crit Care. 2011 Oct;26(5):502-509. doi: 10.1016/j.jcrc.2010.12.015. Epub 2011 Mar 3. PMID 21376523
- [Background] Levy SD, Alladina JW, Hibbert KA, Harris RS, Bajwa EK, Hess DR. High-flow oxygen therapy and other inhaled therapies in intensive care units. Lancet. 2016 Apr 30;387(10030):1867-78. doi: 10.1016/S0140-6736(16)30245-8. Epub 2016 Apr 28. PMID 27203510
- [Background] Sim MA, Dean P, Kinsella J, Black R, Carter R, Hughes M. Performance of oxygen delivery devices when the breathing pattern of respiratory failure is simulated. Anaesthesia. 2008 Sep;63(9):938-40. doi: 10.1111/j.1365-2044.2008.05536.x. Epub 2008 Jun 6. PMID 18540928
- [Background] Roca O, Hernandez G, Diaz-Lobato S, Carratala JM, Gutierrez RM, Masclans JR; Spanish Multidisciplinary Group of High Flow Supportive Therapy in Adults (HiSpaFlow). Current evidence for the effectiveness of heated and humidified high flow nasal cannula supportive therapy in adult patients with respiratory failure. Crit Care. 2016 Apr 28;20(1):109. doi: 10.1186/s13054-016-1263-z. PMID 27121707
- [Background] Parke RL, McGuinness SP. Pressures delivered by nasal high flow oxygen during all phases of the respiratory cycle. Respir Care. 2013 Oct;58(10):1621-4. doi: 10.4187/respcare.02358. Epub 2013 Mar 19. PMID 23513246
- [Background] Frat JP, Thille AW, Mercat A, Girault C, Ragot S, Perbet S, Prat G, Boulain T, Morawiec E, Cottereau A, Devaquet J, Nseir S, Razazi K, Mira JP, Argaud L, Chakarian JC, Ricard JD, Wittebole X, Chevalier S, Herbland A, Fartoukh M, Constantin JM, Tonnelier JM, Pierrot M, Mathonnet A, Beduneau G, Deletage-Metreau C, Richard JC, Brochard L, Robert R; FLORALI Study Group; REVA Network. High-flow oxygen through nasal cannula in acute hypoxemic respiratory failure. N Engl J Med. 2015 Jun 4;372(23):2185-96. doi: 10.1056/NEJMoa1503326. Epub 2015 May 17. PMID 25981908
- [Background] Maggiore SM, Idone FA, Vaschetto R, Festa R, Cataldo A, Antonicelli F, Montini L, De Gaetano A, Navalesi P, Antonelli M. Nasal high-flow versus Venturi mask oxygen therapy after extubation. Effects on oxygenation, comfort, and clinical outcome. Am J Respir Crit Care Med. 2014 Aug 1;190(3):282-8. doi: 10.1164/rccm.201402-0364OC. PMID 25003980
- [Background] Huang HW, Sun XM, Shi ZH, Chen GQ, Chen L, Friedrich JO, Zhou JX. Effect of High-Flow Nasal Cannula Oxygen Therapy Versus Conventional Oxygen Therapy and Noninvasive Ventilation on Reintubation Rate in Adult Patients After Extubation: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. J Intensive Care Med. 2018 Nov;33(11):609-623. doi: 10.1177/0885066617705118. Epub 2017 Apr 21. PMID 28429603
- [Background] Thille AW, Muller G, Gacouin A, Coudroy R, Decavele M, Sonneville R, Beloncle F, Girault C, Dangers L, Lautrette A, Cabasson S, Rouze A, Vivier E, Le Meur A, Ricard JD, Razazi K, Barberet G, Lebert C, Ehrmann S, Sabatier C, Bourenne J, Pradel G, Bailly P, Terzi N, Dellamonica J, Lacave G, Danin PE, Nanadoumgar H, Gibelin A, Zanre L, Deye N, Demoule A, Maamar A, Nay MA, Robert R, Ragot S, Frat JP; HIGH-WEAN Study Group and the REVA Research Network. Effect of Postextubation High-Flow Nasal Oxygen With Noninvasive Ventilation vs High-Flow Nasal Oxygen Alone on Reintubation Among Patients at High Risk of Extubation Failure: A Randomized Clinical Trial. JAMA. 2019 Oct 15;322(15):1465-1475. doi: 10.1001/jama.2019.14901. PMID 31577036
- [Background] Soummer A, Perbet S, Brisson H, Arbelot C, Constantin JM, Lu Q, Rouby JJ; Lung Ultrasound Study Group. Ultrasound assessment of lung aeration loss during a successful weaning trial predicts postextubation distress*. Crit Care Med. 2012 Jul;40(7):2064-72. doi: 10.1097/CCM.0b013e31824e68ae. PMID 22584759
- [Background] Bikker IG, Leonhardt S, Reis Miranda D, Bakker J, Gommers D. Bedside measurement of changes in lung impedance to monitor alveolar ventilation in dependent and non-dependent parts by electrical impedance tomography during a positive end-expiratory pressure trial in mechanically ventilated intensive care unit patients. Crit Care. 2010;14(3):R100. doi: 10.1186/cc9036. Epub 2010 May 30. PMID 20509966
- [Background] Wang G, Zhang L, Li B, Niu B, Jiang J, Li D, Yue Z, Weng Y. The Application of Electrical Impedance Tomography During the Ventilator Weaning Process. Int J Gen Med. 2021 Oct 16;14:6875-6883. doi: 10.2147/IJGM.S331772. eCollection 2021. PMID 34703292
- [Background] Hughes, Martin, and Roland Black (eds), Advanced Respiratory Critical Care, Oxford Specialist Handbooks (Oxford, 2011; online edn, Oxford Academic, 1 Oct. 2011), https://doi.org/10.1093/med/9780199569281.001.0001, accessed 5 May 2023.